CLINICAL TRIAL: NCT00102375
Title: Phase III Multicenter Study in Epithelial Ovarian Carcinoma FIGO Stage IIB-IV Comparing Treatment With Paclitaxel and Carboplatin to Paclitaxel and Carboplatin Sequentially Followed by Topotecan
Brief Title: Paclitaxel, Carboplatin, and Topotecan in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 7
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; first-line; Topotecan
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
The purpose of this study is to determine whether the triple combination of Carboplatin, Paclitaxel and Topotecan has a superior clinical outcome in the treatment of ovarian cancer compared with the combination of Carboplatin and Paclitaxel.

DETAILED DESCRIPTION:
Carboplatin-Paclitaxel is the current standard in the first-line treatment of advanced ovarian cancer. One option to further improve the therapeutic results is the incorporation of a third, non-cross-resistant drug into first line chemotherapy of advanced ovarian cancer. In two separate, single center phase II studies, a different combination of the three active agents (Carboplatin, Paclitaxel and Topotecan) has been tested. In these studies, Carboplatin and Paclitaxel were given at standard doses and schedules, followed sequentially by Topotecan which was well tolerated at a dose of 1.25 mg/m2/day given for five days and repeated every 21 days. The prolonged therapy is not associated with cumulative toxicity and the compliance of the patients was good.

Study Hypothesis/Comparison: The triple combination (Carboplatin/Paclitaxel/Topotecan) yields superior outcome in the treatment of first-line ovarian cancer compared with the combination of Carboplatin + Paclitaxel

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epithelial carcinoma of the ovary or of the fallopian tube or extraovarian papillary serous carcinoma with extent to the ovary
* International Federation of Gynecology and Obstetrics (FIGO) stage IIB-IV, regardless of measurable or non-measurable disease
* No prior chemo- or radiotherapy
* Adequate hematologic, renal and hepatic function:

  * ANC ≥ 1.5 x 10^9/L,
  * Platelet counts ≥ 100 x 10^9/L,
  * Total bilirubin ≤ 1.5 x upper normal limit,
  * Alkaline Phosphatase ≤ 3 x upper normal limit,
  * Serum creatinine ≤ 1.25 upper normal limit,
  * Estimated GFR ≥ 60 ml/min
* Performance status 0-2 (ECOG)
* Life expectancy must be greater than 12 weeks

Exclusion Criteria:

* Non-epithelial tumors or mixed epithelial/non-epithelial tumors (e.g. mixed Mullerian tumors) or tumors of low malignant potential (borderline tumors)
* Prior treatment with chemo- or radiotherapy
* Administration of other simultaneous chemotherapeutic drugs or hormonal therapy or simultaneous radiotherapy during the study treatment period or planned whole abdominal radiotherapy
* History of congestive heart failure
* Symptomatic brain metastasis
* Complete bowel obstruction
* Dementia
* Active infection or other serious underlying medical condition
* Pre-existing motor or sensory neurologic pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 1999-12; Study Completion 2004-10

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Progression-free survival
Response rate
Response duration
Toxicities
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, Prof. Dr., Principal Investigator — AGO Study Group
Locations (18):
- Germany (18):
  - Gynecologic Hospital of the Medical Facilities RWTH, Aachen
  - Clinic for Gynecology and Gyn. Oncology, Humboldt University, Berlin
  - University Clinic Carl Gustav Carus, Gynecological hospital, Dresden
  - Gynecologic Hospital, Düsseldorf
  - University Gynecologic Hospital, Düsseldorf
  - University Gynecologic Hospital, Frankfurt
  - University Gynecologic Hospital, Göttingen
  - Gynecologic Clinic of the Ernst-Moritz-Arndt-University, Greifswald
  - Gynecological Clinic of the Medical University, Hanover
  - St. Vincentius Gynecologic Hospital, Karlsruhe
  - University Clinic Schleswig-Holstein, Campus Kiel, Clinic for gynecology and obstetrics, Kiel
  - Otto-von-Guericke University, University Gynecological Hospital, Magdeburg
  - University Gynecologic Hospital Grosshadern, München
  - University Gynecologic Hospital "rechts der Isar", München
  - Clinic for Gynecology, Münster
  - University Gynecologic Hospital, Tübingen
  - University Gynecological Hospital, Ulm
  - Clinic for Gnyecology and gyn. Oncology HSK, Wiesbaden

REFERENCES:
- [Result] Pfisterer J, Weber B, Reuss A, Kimmig R, du Bois A, Wagner U, Bourgeois H, Meier W, Costa S, Blohmer JU, Lortholary A, Olbricht S, Stahle A, Jackisch C, Hardy-Bessard AC, Mobus V, Quaas J, Richter B, Schroder W, Geay JF, Luck HJ, Kuhn W, Meden H, Nitz U, Pujade-Lauraine E; AGO-OVAR; GINECO. Randomized phase III trial of topotecan following carboplatin and paclitaxel in first-line treatment of advanced ovarian cancer: a gynecologic cancer intergroup trial of the AGO-OVAR and GINECO. J Natl Cancer Inst. 2006 Aug 2;98(15):1036-45. doi: 10.1093/jnci/djj296. PMID 16882940
- See also: Information on studies of the AGO-OVAR on Ovarian cancer — http://www.ago-ovar.de